CLINICAL TRIAL: NCT00039689
Title: Leukapheresis Procedures to Obtain Plasma and Lymphocytes for Research Studies on Antiretroviral Naive HIV-1 Research Participants
Status: Recruiting | Type: Observational
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 020202; 02-I-0202
Record Dates: First submitted 2002-06-06; First posted 2002-06-07 (Estimated); Last update posted 2026-01-16 (Actual); Status verified 2025-07-07

CONDITIONS: HIV
Keywords: Cellular Immunity; Chronic HIV Infection; Antiretroviral Therapy; Primary HIV Infection; Humoral Immunity; Natural History; HIV Infection; Acute Infection; Treatment Naive
MeSH Terms: conditions — HIV Infections

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- HIV chronic infection: For example, an individual infected with HIV-1 for an indeterminate amount of time.
- HIV early infection: For example, a negative HIV antibody immunoassay within 6 months of a positive HIV antibody assay and confirmatory test (as defined by current CDC criteria).

SUMMARY:
There is evidence that early and aggressive treatment with antiretroviral drugs can prevent the loss of immune cell function that accompanies HIV infection. This study will use leukapheresis (drawing blood, separating out the white cells and returning the blood to the patient) to obtain blood cells from HIV-infected patients in either the acute or chronic stage of infection who are being treated with early highly active antiretroviral therapy (HAART). Leukapheresis is necessary to obtain enough cells to delineate the response of B cells to CD4+ T cell help, the CD8 factors associated with suppression of viral replication and normalization of immune function, and natural killer function relative to HIV disease.

Study participants will be adult (older than 18 years) HIV primary or acutely affected patients (those with a history of exposure to HIV but not yet showing chronic symptoms of HIV disease) and HIV chronically infected patients (those infected with HIV for longer than 12 months or showing other symptoms of HIV disease) who are not receiving HAART at the beginning of the study. The study seeks to enroll 30 primary and 30 chronic patients. Pregnant women will not be enrolled in the study; women who become pregnant will be dropped from the study.

Leukapheresis will be performed on each patient before HAART therapy begins and then three times a year. Each session will take between 1 and 3 hours.

This longitudinal study will enable researchers to examine the function of certain B cells, natural killer cells, and CD8+ T cells in people who do not have chronic HIV disease and in those who do have the disease and are treated with HAART.

...

DETAILED DESCRIPTION:
HIV-1 infection is known to cause profound and irreversible dysfunction of both innate and adaptive arms of the immune system. However, there is mounting evidence that early and aggressive treatment with antiretroviral drugs can prevent loss of immune cell function. In an attempt to further delineate the effect of early antiretroviral therapy (ART) on maintenance of immune cell function, we wish to recruit people with drug-naive HIV-1 who are either in early or chronic stage of the disease. The study will require that participants undergo leukapheresis or research blood draw once before and several times after enrollment. Leukapheresis will be used in order to obtain sufficient cells to pursue the following objectives: delineating B cell response to CD4+ T cell help, delineating the effect of ART on persistent HIV reservoirs in CD4+ T cells of people with HIV (PWH), and delineating CD8+ T cell-mediated suppression of viral replication and normalization of immune function, and characterizing natural killer (NK) function relative to HIV disease. The required number of mononuclear cells needed to perform these experiments can be easily and safely obtained using leukapheresis procedures in the Clinical Center Apheresis Unit. This protocol is specifically designed to conform to the requirements of the Apheresis Unit for donors to have leukapheresis procedures, but the protocol, by itself, is not an independent research study. Alternatively, whole blood draws may be used in cases where participants are unable to undergo leukapheresis. While this approach will limit extensive functional analyses, informative phenotypic and limited functional analyses can nonetheless be performed.

ELIGIBILITY:
* INCLUSION CRITERIA:

  1. Adult (18 years old or older) with HIV-1.
  2. Adequate venous access for research blood collection.
  3. Positive HIV antibody immunoassay and a positive confirmatory HIV test (as defined by current CDC criteria). Tests may be done in our clinic or by an outside provider. For individuals with suspected early HIV-1, the following additional criteria may be used: HIV-1 RNA levels of >2,000 copies/ml with a negative result from an HIV antibody immunoassay.
  4. Willingness to be able to make follow up visits at least once in the next 4 months and prior to the initiation of antiretroviral therapy (ART).
  5. Blood pressure < 180/100; pulse rate between 50-100 unless a lower pulse rate is considered normal for the volunteer.
  6. Adequate blood counts (hemoglobin greater than or equal to 9.0 g/dL, hematocrit greater than or equal to 28 percent, platelets greaterhan or equal to 50,000).
  7. Willingness and ability to give informed consent including consent for the storage of blood samples and genetic testing.
  8. Antiretroviral naive, no antiretroviral use in the last six months, or previously enrolled 02-I-0202 participants on whom there are samples stored in the repository.

     1. Participants who acquire HIV-1 while taking ART for pre-exposure prophylaxis will be eligible for enrollment as long as they meet diagnostic criteria for HIV positivity.
     2. Participants who enroll under another LIR apheresis protocol within the past three months and complete the apheresis within 4 weeks of starting ART will also be eligible for enrollment.
     3. Participants with limited (no more than 4 weeks before screening visit) recent use of ART may be eligible for study participation if, the opinion of the investigator, the ART usage will not impact the scientific validity of the protocol.

EXCLUSION CRITERIA:

1. Pregnant and / or breastfeeding.
2. Be currently abusing alcohol or other drugs that potentially could interfere with the participant s compliance or safety.
3. Have a condition which in the opinion of the investigators would make the participant ineligible for the study.

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants will be recruited from existing cohorts of individuals participating in National Institute of Allergy and Infectious Diseases (NIAID) who meet the Inclusion/Exclusion Criteria. Additional local and regional recruitment may be done using direct mailing to infectious disease physicians, internet ad campaigns, social media outlets, print ads, and from local clinics via the NIAID patient recruitment contract with Matthews Media Group.
Sampling Method: Non-Probability Sample
Enrollment: 750 (Estimated)
Dates: Start 2002-07-12 (Actual)

PRIMARY OUTCOMES:
To further investigate differences in the immunologic function of various lymphocyte subsets in PWH who are treated early after transmission of HIV and during the chronic phase of the disease. | Throughout the study
  To further investigate differences in the immunologic function of various lymphocyte subsets in PWH who are treated early after transmission of HIV and during the chronic phase of the disease. Studies will also be done to further delineate the various antigen-specific and innate immune responses including characterization of soluble factors associated with early HIV disease.

CONTACTS AND LOCATIONS:
Overall Officials: Susan L Moir, Ph.D., Principal Investigator — National Institute of Allergy and Infectious Diseases (NIAID)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

REFERENCES:
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?A_2002-I-0202.html